CLINICAL TRIAL: NCT01793558
Title: Study That Evaluates the Incidence and Possibilities for Prevention of Hypothermia in Newborns Bonding During Caesarean Section
Brief Title: Incidence and Prevention of Hypothermia in Newborns Bonding During Caesarean Section
Acronym: THER5
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, PD Dr. Jan Hoecker, Associate Professor of Anaesthesiology, University Hospital Schleswig-Holstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THER-5
Record Dates: First submitted 2013-02-12; First posted 2013-02-15 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Thermoregulation Impairment; Hypothermia; Postoperative Shivering
Keywords: Thermoregulation Impairment; hypothermia; Postoperative shivering; cesarean section; newborn
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control; passive insulation (No Intervention): The mothers will receive passive temperature insulation by a cotton blanket (standard procedure) after start of the spinal anaesthesia for cesarean section. The newborn will be bonded on the mothers chest under the cotton blanket (also passive insulation without active warming) for 20 min after birth (bonding period).
- Active Warming (Experimental): The mothers will receive active warming by a forced-air warming blanket after start of the spinal anaesthesia for cesarean section. The newborn will be bonded on the mothers chest under the warming blanket for 20 min after birth (bonding period).
  Interventions: Procedure: Forced-air warming

INTERVENTIONS:
Procedure: Forced-air warming — In the intervention group a forced-air cover (Level 1 Snuggle Warm Upper Body Blanket, Smiths Medicals) will be positioned over the upper body of the patients laying on the operating table just beginning after the spinal block.
  Other Names: Level 1 Snuggle Warm Upper Body Blanket; Forced-air warming blower
  Arms: Active Warming

SUMMARY:
This study should evaluate whether newborns during cesarean section are endangered to get hypothermic while bonding on the mothers chest.

Therefore, the investigators want to investigate the effects of active cutaneous warming of the mothers and babies during intraoperative bonding. The investigators plan to enroll 40 parturients scheduled for elective caesarean section to receive passive insulation or forced-air skin surface warming. The investigators will measure core temperature of the newborns and their mothers. The investigators hypothesize that newborns became most often hypothermic without active warming during the bonding procedure and that active warming will be able to decrease the number of hypothermic newborns significantly.

DETAILED DESCRIPTION:
Little is known about the thermoregulatory effects on babies when bonding on the chest of the mother during caesarian section. The aim of our study is to evaluate whether newborns during cesarean section are endangered to get hypothermic while bonding on the mothers chest. The investigators want to investigate the effects of active cutaneous warming of the mothers and babies during a 20 min intraoperative bonding period. The investigators plan to enroll 40 parturients scheduled for elective caesarean section under spinal anaesthesia to receive passive insulation or forced-air skin surface warming. The investigators will measure core temperature of the newborns and their mothers. The investigators hypothesize that newborns became most often hypothermic without active warming during the bonding procedure and that active warming will be able to decrease the number of hypothermic newborns significantly.

ELIGIBILITY:
Inclusion Criteria:

* parturients undergoing planned, elective cesarean section under spinal anaesthesia
* mothers classified as American Society of Anaesthesiologists (ASA) status I or II
* written informed consent

Exclusion Criteria:

* mothers younger than 18 years
* mothers classified as American Society of Anaesthesiologists (ASA) status III or higher
* caesarean section planned under general anaesthesia.
* any expected problems with the newborn such as:

  * gestation date < 36 or > 42 week
  * placenta previa, abruption of placenta, green amniotic fluid, amnion infection syndrome or any abnormalities in cardiotocography (CTG)

Max Age: 20 Minutes | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2013-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Body core temperature of the newborn | 20 min after birth
  Core temperature of the infants will be measured with specific probes 20 min after birth (end of bonding period)by a rectal temperature probe.

SECONDARY OUTCOMES:
Skin temperature of the newborn | 20 min after child birth
  Skin temperature of the infants will be measured with specific probes 20 min after birth (end of bonding period) at chest, arm, thigh, and calf. Mean-skin temperature will be calculated from these measurements.

OTHER OUTCOMES:
Shivering incidence of the mothers | 20 min after child birth
  Shivering of the mothers will be graded by a four-point scale.
Thermal comfort of the mothers | 20 min after child birth
  Thermal comfort of the mother will be evaluated with a 100-mm visual analogue scale.
Mean arterial blood pressure of the mothers. | 20 min after child birth
  Mean arterial blood pressure of the mothers will be assessed by non-invasive measurement.
Core temperature of the mothers | 20 min after child birth
  Core temperature will be measured by a sublingual temperature probe.
Skin temperature of the mothers. | 20 min after child birth
  Skin temperature of the mothers will be assessed at the chest.

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Bein, M.D., Study Chair — University Hospital Schleswig-Holstein, Campus Kiel, Kiel, Germany
Locations (1):
- Klinikum Pinneberg Klinik für Anästhesiologie, Intensivmedizin und OP-Management, Pinneberg, Schleswig-Holstein, Germany